CLINICAL TRIAL: NCT03249818
Title: Feasibility Study of Head and Intraocular Trauma Test (HITT) Device for Potential Detection of Brain Dysfunction
Brief Title: HITT Device Pilot Testing for Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rebiscan, Inc. (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: rebiscan-004
Record Dates: First submitted 2017-08-09; First posted 2017-08-15 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- HITT Device (Other): HITT device to scan eyes of participants 3 times (30 seconds each) at time of admittance to hospital for diagnosed traumatic brain injury. If patient is still in hospital 2 weeks post-enrollment, a second set of 3 tests will be performed
  Interventions: Device: HITT device

INTERVENTIONS:
Device: HITT device — Device scans the fovea of the eye to measure fixation. Patients will then be asked to track the fixation target across an area the size of a playing card, with the device tracking the participant's fixation throughout.

SUMMARY:
The purpose of this research study is to collect data from the eyes of traumatic brain injury (TBI) patients. Patients will look at a green target that will measure the fixation of the eye for 30 seconds. In that 30 seconds, the location of the green target will change and the participant is to track, with their eyes, the light as best they can. The device will measure how well fixation was maintained and the speed of the saccadic movements of the eye. Data will then be used to determine whether there is correlation between these measures and known TBI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18-40
2. Documented/ verified mild TBI
3. Mild traumatic brain injury will be defined as Glasgow Coma Scale (GCS) of ≥13 at time of study enrollment
4. Injury occurred < 24 hours ago
5. Positive acute brain CT for clinical care
6. Visual acuity/ hearing adequate for testing
7. Fluency in English or Spanish
8. Ability to provide informed consent
9. Enrolled in TRACK-TBI (IRB #: 825503)

Exclusion Criteria:

1. Catastrophic polytrauma that would interfere with follow-up and outcome assessment
2. Prisoners or patients in custody
3. Pregnancy in female subjects
4. Patients on psychiatric hold (e.g. 5150, 5250)
5. Major debilitating baseline mental health disorders (e.g. schizophrenia or bipolar disorder) that would interfere with follow-up and the validity of outcome assessment
6. Major debilitating neurological disease (e.g. stroke, dementia, tumor) impairing baseline awareness, cognition, or validity of follow-up and outcome assessment
7. Significant history of pre-existing conditions that would interfere with follow-up and outcome assessment (e.g. substance abuse, alcoholism, HIV/AIDS, major transmittable diseases that may interfere with consent, end-stage cancers, learning disabilities, developmental disorders)
8. Low likelihood of follow-up (e.g. participant or family indicating low interest, homelessness or lack of reliable contacts)
9. Penetrating TBI
10. Spinal cord injury with ASIA (American Spinal Injury Assoc.) score of C or worse
11. Any injury to eye including, puncture, scratch, occlusion, fracture to orbital socket (or any fracture to face that would negatively impact eye movement/vision) that would interfere with ability to complete study-device assessment.
12. History of poor vision prior to injury (Visual acuity worse than 20/40 in either eye)
13. Intoxication or chemical impairment at time of examination (upon initial presentation)
14. Evidence on hand-light examination of obvious ocular anomaly or misalignment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
TBI detection | 1 day
  Patients who have diagnosed TBI and are admitted to the hospital for treatment will have their eyes scanned to identify whether the HITT device can accurately identify patients with TBI

SECONDARY OUTCOMES:
TBI monitor | 14 days
  Patients who have remained in the hospital for TBI and received initial HITT device scan will receive a second set of scans at 2 weeks to identify whether the HITT device can accurately identify patients with TBI

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Diaz-Arrastia, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregate data and individual test reports will be made available to the HITT device manufacturer to better understand its performance at identifying TBI. Personal identifiable data will not be shared with anyone outside of the University of Pennsylvania.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be shared on an ongoing basis, and cumulatively at the end of the study. Study length is expected to be 2 months from first enrolled participant.
Access Criteria: Data will only be shared with researchers involved in the study at the University of Pennsylvania, and only trained staff members at the device manufacturer.